CLINICAL TRIAL: NCT04093856
Title: Determinants of Bone and Muscle Quality and Strength in Obesity With and Without Diabetes
Acronym: BODI2
Status: Completed | Type: Observational
Sponsor: Suzanne Morin (Other)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor-Investigator, Suzanne Morin, Clinician Researcher, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: MP-37-2020-5872
Record Dates: First submitted 2019-09-10; First posted 2019-09-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity; Body Weight; Bone Diseases, Metabolic; Fractures, Bone; Osteoporotic Fractures; Osteoporosis; Quality of Life; Fall; Musculoskeletal Diseases
Keywords: Advanced glycation end products; Advanced imaging; Mobility; Strength
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity; Body Weight; Bone Diseases, Metabolic; Fractures, Bone; Osteoporotic Fractures; Osteoporosis; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic: 20 men and women with type 2 diabetes and obesity
- Non-diabetic: 20 normoglycemic men and women with obesity matched for age and sex with diabetic group

SUMMARY:
Background: Osteoporotic fractures are a major public health issue. They cause substantial disability, loss of autonomy, morbidity and excess mortality. Diabetes is also associated with increased risk for falls and fractures through a direct impact of elevated blood glucose on the skeleton and on muscles.

Research project overview: The investigators propose a cross-sectional study that will involve 2 research centers in the province of Quebec. The investigators will recruit 20 obese participants, without diabetes, who have not undergone bariatric surgery, for one-time measurements to be compared with baseline measurements (pre-surgery) from participants in the bariatric obese diabetic groups with type II diabetes mellitus from the ongoing study BODI study (NCT03455868). Bone Mineral Density as well as muscle quality, strength and function will be evaluated at a single study visit.

Relevance: This data will permit the evaluation of the bone-muscle unit in patients with obesity with and without diabetes, and assess whether the presence and duration of diabetes impacts further on clinical and functional musculoskeletal outcomes (falls, fractures and mobility and strength) in this population. AGEs, if associated with muscle and bone deterioration, might become an easily accessible biomarker of musculoskeletal health in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

A) Diabetic group

* BMI >=35 kg/m2
* Clinical diagnosis of type 2 diabetes
* Use of oral hypoglycemic agents or insulin or 2 of the following tests confirming type 2 diabetes: HbA1c >=6.5%; fasting glucose >=7.0 mM; 2-h glucose post 75g oral glucose tolerance test (OGTT) >=11.1 mM)

B) Non-diabetic group:

* BMI >=35 kg/m2
* Normoglycemia (HgbA1c <5.7% and Fasting glucose <5.6 nM)

Exclusion Criteria:

* BMI >60 kg/m2
* Clinical diagnosis of type 1 diabetes
* Disease (e.g. uncontrolled thyroid disease, malabsorptive or overt inflammatory disorder, metabolic bone disease, creatinine clearance <60 ml/min)
* Medication (e.g. gluccocorticoids, anti-epileptic drugs, osteoporosis therapy and thiazolidinediones) affecting bone metabolism
* Pregnancy
* History of oesophageal, gastric, digestive or bariatric surgery
* Prosthesis that could interfere with interpretation of imaging data
* Chronic severe condition or illness precluding from participation in the project.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a multi-center, cross-sectional, observational study comprising of two groups of participants with obesity either with or without diabetes (n=20/group). The diabetic groups will include 20 adult men and women with obesity and type 2 diabetes, and the non-diabetic group will consist of 20 age- and sex- matched individuals with obesity and normoglycemia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Muscle size measured as cross-sectional muscle area at the proximal femur | Baseline
  Measured by quantitative computed tomography (QCT)
Muscle composition measured as muscle fat content at the proximal femur | Baseline
  Measured by quantitative computed tomography (QCT)
Volumetric bone mineral density (vBMD) at the spine, hip, radius and tibia | Baseline
  Measured by quantitative computed tomography (QCT)

SECONDARY OUTCOMES:
N-terminal propeptide of type 1 procollagen concentration | Baseline
  Serum bone formation marker
Osteocalcin (total and decarboxylated) concentration | Baseline
  Serum bone formation marker
Bone specific alkaline phosphatase concentration | Baseline
  Serum bone formation marker
C-telopeptide concentration | Baseline
  Serum bone resorption marker
Fasting glucose concentration | Baseline
  Diabetes control
Fasting Hemoglobin A1c concentration | Baseline
  Diabetes control
Insulin concentration | Baseline
  Hormone involved in bone metabolism
Serum 25-hydroxyvitamin D concentration | Baseline
  Hormone involved in bone metabolism
Parathormone concentration | Baseline
  Hormone involved in bone metabolism
Estradiol concentration | Baseline
  Hormone involved in bone metabolism
Insulin like growth factor-1 concentration | Baseline
  Hormone involved in bone metabolism
Sclerostin concentration | Baseline
  Hormone involved in bone metabolism
Adiponectin concentration | Baseline
  Hormone involved in bone metabolism
Leptin concentration | Baseline
  Hormone involved in bone metabolism
Body composition measured as visceral and subcutaneous adipose tissue | Baseline
  Measured by computed tomography (CT)
Body composition measured by fat and lean mass | Baseline
  Measured using dual-energy X-ray absorptiometry (DXA)
Bone marrow adiposity | Baseline
  Measured by computed tomography (CT)
Upper extremity muscle strength measured by grip force in kg | Baseline
  Measured using Jamar Hydraulic Hand Dynamometer
Lower extremity muscle strength measured by peak torque generated by knee extension | Baseline
  Measured using Biodex isokinetic dynamometer
Functional mobility measured by time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. | Baseline
  Measured using Timed Up and Go test.
Functional exercise capacity measured by total distance ambulated during a 6 minute time period | Baseline
  Measured using Six Minute Walk Test
Self-reported physical activity measured in metabolic equivalents (MET) | Baseline
  Measured using the International Physical Activity Questionnaire
Cutaneous Advanced glycation end products (AGEs) measurement | Baseline
  Measured by measured by AGE Reader
Physical activity measured by total activity and time spent in different intensities of exercise measured over 7 consecutive days | Baseline
  Actigraph GT3X+ Accelerometer
Functional balance score obtained using multidimensional balance assessment. Higher scores indicate better balance abilities | Baseline
  Fullerton Advanced Balance (FAB) Scale
Physical health | Baseline
  SF-12
Community Participation Restriction | Baseline
  Life-space mobility assessment
Health-related quality of life | Baseline
  How are you today? Visual analogue scale

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Centre de recherche de l'IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: No